CLINICAL TRIAL: NCT06255470
Title: Effect of Periodontal Treatment on Salivary and Serum SIRT-1, MMP-9 and T-SOD Levels
Brief Title: Effect of Periodontal Treatment on Salivary and Serum Biomarkers in Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.2022.863
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Periodontal Health; Periodontitis
Keywords: periodontitis; periodontal treatment
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Periodontally Healthy (No Intervention): Periodontally healthy patients received no intervention.
- Periodontitis Stage III Grade B (Active Comparator): The patients were subjected to quadrant-wise full-mouth subgingival scaling and root planning under local anesthesia by the use of ultrasonic scalers and curettes. The entire non-surgical periodontal treatment of periodontitis groups was completed in a total of 4 sessions in two weeks.
  Interventions: Procedure: Non-surgical periodontal treatment
- Periodontitis Stage III Grade C (Active Comparator): The patients were subjected to quadrant-wise full-mouth subgingival scaling and root planning under local anesthesia by the use of ultrasonic scalers and curettes. The entire non-surgical periodontal treatment of periodontitis groups was completed in a total of 4 sessions in two weeks.
  Interventions: Procedure: Non-surgical periodontal treatment

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Non-surgical periodontal treatment involves the removal of microbial dental plaque and calculus by mechanical debridement using manual and ultrasonic instruments. Motivating and educating patients about oral hygiene procedures is another important part of the treatment. The aim is to stop the progression of the disease and to prevent the occurrence of active clinical inflammation.
  Arms: Periodontitis Stage III Grade B; Periodontitis Stage III Grade C

SUMMARY:
The present study aimed to determine the effect of non-surgical periodontal treatment on serum and salivary SIRT-1, MMP-9, and T-SOD levels in periodontitis stage III grade B (P-III-B) and C (P-III-C) patients. 17 periodontally healthy, 16 P-III-B and 16 P-III-C subjects were enrolled. At baseline, serum and saliva samples were collected and the whole mouth clinical periodontal parameters were recorded. Periodontitis patients received non-surgical periodontal treatment. Clinical parameters were re-measured and samples were re-collected at 3 months after treatment. Serum and salivary SIRT-1, MMP-9, and T-SOD levels were analyzed by ELISA. Data were analyzed using appropriate statistical tests.

DETAILED DESCRIPTION:
Periodontitis is a dysbiotic chronic inflammatory disease that compromises the integrity of the tooth-supporting tissues. When periodontitis occurs, reactive oxygen species, which are overproduced mostly by hyperactive neutrophils, can not be balanced by the antioxidant defense system and cause tissue damage. Cytoprotective enzymes such as superoxide dismutase (SOD), catalase (Cat) and the regulatory pathways that influence them, play a critical role in the scavenging and detoxification of ROS. Sirtuin-1 (SIRT-1) is a nicotinamide adenine dinucleotide (NAD)dependent histone deacetylase. SIRT1 is known to deacetylate FOXO3a, which induces antioxidant responses via modulation in SOD2 and CAT. Moreover, SIRT1 overexpression downregulates the pro-inflammatory cytokines such as interleukin (IL)-1α, IL-6, IL-8 and tumor necrosis factor-α (TNF-α) synthesis which are associated with the onset and progression of the periodontal disease. MMP-9 is a host-derived proteolytic enzyme that leads to periodontal tissue breakdown and is activated by oxidative stress.

This study aims to examine the effect of non-surgical periodontal treatment (NSPT) on saliva and serum SIRT-1, SOD and MMP-9. It is the first controlled clinical study investigating the effect of NSPT on salivary SIRT-1 levels in different periodontitis groups. The sample size was calculated based on a previous study investigating the level of salivary MMP-9 and the power of the test was 95%, alfa value: 0.05. The estimated sample size was 10 individuals for each group. Therefore, a total of 49 systemically healthy patients; 17 periodontally healthy, 16 P-III-B, 16 P-III-C were included in this study. Periodontal examination was performed, and full medical and dental histories were collected by a single examiner at baseline and 3 months after NSPT. The whole mouth clinical periodontal examination included measurement of probing depth (PPD), clinical attachment level (CAL), presence of bleeding on probing (BOP), gingival index (GI), and plaque index (PI) at 6 sites per tooth, except the third molars. The presence and type of the alveolar bone loss were assessed on the digital panoramic radiograph in each participant, which was supplemented with periapical radiographs if necessary. Periodontal status of each patient was evaluated by a single calibrated periodontists with a manual probe. The diagnosis of periodontitis or periodontal health was determined according to the 2017 World Workshop on Classification of Periodontal and Peri-Implant Diseases and Conditions. Periodontally healthy individuals (n=17) in the control group had no sites with PD >3 mm and CAL >2 mm and also no radiographic evidence of alveolar bone loss. BOP was <10%.

The periodontitis stage III patients had a minimum of three teeth apart from the first molars and incisors showing CAL ≥5 mm and PD ≥6 mm and showed no>4 teeth loss because of periodontitis. Radiographic bone loss extending from coronal to middle third or beyond. Radiographic bone loss was determined from the tooth showing the most severe bone loss as a percentage of root length. If the values of bone loss %/age were between 0.25 and 1.0, the patients were assigned to grade B (n=16). If higher than 1.0, the patients were assigned to grade C (n=16).

Treatment

Patients in the periodontitis groups underwent quadrant-wise supra and subgingival mechanical scaling and root planing using ultrasonic scalers and manual instruments, after administration of local anesthesia. No periodontal intervention was carried out in the periodontally healthy controls.

Saliva and Serum Sampling

A total of 5 mL of unstimulated whole saliva was collected by passive drool method between 9:00 and 10:00 am. The participants were advised to avoid food consumption for three hours before sample collection. The participants were seated upright, and saliva was collected over a period of 5 minutes with instructions to pool saliva in the floor of the mouth and passively drool it into a sterile glass beaker. Then saliva samples are immediately transferred to a 2 mL polypropylene tube and stored at -80°C. A total of 5 mL of blood was collected from the antecubital fossa by vene puncture method. Serum was isolated from the blood by centrifuging at 5000 rpm for 10 minutes followed by its rapid transfer to a sterile polypropylene tube and storage at -80°C.

Biomarker Immunoassays Saliva and serum samples were thawed on ice. The saliva samples were centrifuged at 5.000 rpm for 15 minutes at room temperature, and supernatants were immediately used for assays. Serum and salivary samples of SIRT-1 , MMP-9, MIP-1α*, T-SOD were measured by ELISA using commercial kits.

Statistical Analysis

All statistical analyses were carried out with the standard statistical software package. For the intra-group comparisons, if the data were not normally distributed, Wilcoxon-signed rank test and the Dunn test with the Bonferroni correction were used to analyze the change between baseline and 3 months after treatment. For inter-group comparisons, Mann-Whitney U test for normally and non-normally distributed data. The Spearman's rank correlation test was used to detect the correlations of biochemical parameters with clinical parameters and each other's in diseased group before and after treatment. All tests were performed at significance level of P <0.05.

ELIGIBILITY:
Inclusion Criteria:

1. systemically healthy and non-smoker individuals
2. having ≥20 teeth present (except third molars)
3. individuals with periodontally healthy, periodontitis stage III grade B and C diagnoses

Exclusion Criteria:

1. having any diagnosed medical disorders such as diabetes mellitus, cardiovascular diseases, rheumatoid arthritis, immunological and mucocutaneous diseases
2. usage of antibiotics, non-steroidal anti-inflammatory drugs and immunosuppressive agents within the past 6 months
3. having any non-inflammatory destructive periodontal disease
4. nonsurgical/surgical periodontal therapy received in the past year
5. pregnant/ lactating/ postmenopausal females.

Ages: 23 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Salivary SIRT-1 (ng/mL) level | baseline to 3 months after treatment
  change in salivary SIRT-1 levels from baseline to 3 months after treatment
Salivary MMP-9 (ng/mL) level | baseline to 3 months after treatment
  change in salivary MMP-9 levels from baseline to 3 months after treatment
Salivary T-SOD (U/mL) level | baseline to 3 months after treatment
  change in salivary T-SOD levels from baseline to 3 months after treatment

SECONDARY OUTCOMES:
Serum SIRT-1 (ng/mL) level | baseline to 3 months after treatment
  change in serum SIRT-1 levels from baseline to 3 months after treatment
Serum MMP-9 (ng/mL) level | baseline to 3 months after treatment
  change in serum MMP-9 levels from baseline to 3 months after treatment
Serum T-SOD (U/mL) level | baseline to 3 months after treatment
  change in serum T-SOD levels from baseline to 3 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Faculty of Dentistry, Department of Periodontology, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Iyigun S, Gorgulu NG, Dogan B. Changes in MMP-9, T-SOD and SIRT-1 levels after non-surgical periodontal treatment. BMC Oral Health. 2025 Feb 19;25(1):262. doi: 10.1186/s12903-025-05610-5. PMID 39972299